CLINICAL TRIAL: NCT02085057
Title: Shared and Unique Neural Links Between OCD and Anorexia: Investigating Biological Mechanisms of Phenotypic Expression
Brief Title: Neural Links Between OCD and Anorexia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cara Bohon, PhD, Assistant Professor, Stanford University
Other Study IDs: 18888
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Anorexia Nervosa; Obsessive-compulsive Disorder
MeSH Terms: conditions — Anorexia Nervosa; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- anorexia nervosa: Diagnosis of anorexia nervosa
  Interventions: Procedure: Functional Magnetic Resonance Imaging
- obsessive-compulsive disorder: Diagnosis of obsessive-compulsive disorder
  Interventions: Procedure: Functional Magnetic Resonance Imaging
- healthy control: No psychiatric diagnoses
  Interventions: Procedure: Functional Magnetic Resonance Imaging
- sisters: Sisters of those enrolled with a diagnosis of anorexia nervosa
  Interventions: Procedure: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Functional Magnetic Resonance Imaging

SUMMARY:
Individuals with anorexia nervosa (AN) have long been observed to demonstrate symptoms in common with obsessive-compulsive disorder (OCD), in particular, an obsessive fear of normal weight leading to dangerous food restriction, as well as many compulsive rituals about food. Both AN and OCD are seriously handicapping and often resistant to conventional therapies. Given that the two conditions often co-occur and are associated with still unknown genetic risk factors, the aim of this project is to identify their shared and distinct patterns of brain activity.

The investigators propose to use functional magnetic resonance imaging to compare brain response among adolescents with AN, OCD, and age-matched healthy individuals. Specifically, this study will investigate function of distinct brain circuits related to core aspects of these related disorders. The investigators use three tasks related to set shifting, global vs. local processing, and reward. Based on evidence of deficits in cognitive flexibility and ability to change behavior, the investigators hypothesize that adolescents with AN and with OCD will show hypoactivity of frontostriatal circuitry during cognitive tasks, and adolescents with AN will show hyperactivity in limbic regions in a reward task.

This study is the first to directly compare brain activation patterns using functional neuroimaging in AN and OCD. The goal is to determine how abnormal brain activity relates to symptom formation, what accounts for shared characteristics amongst these disorders, and whether deficits in specific circuitry underlie their unique defining features. The study of shared and unique elements of functional brain circuitry reflects a new, emerging approach to the classification of psychiatric illness, one based on identifying unique combinations of biological risk factors that link related conditions. This approach is widely believed to be a critical step forward in developing more brain-relevant targeted strategies for preventative interventions.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 12-19
* anorexia nervosa diagnosis OR obsessive-compulsive diagnosis OR no psychiatric disorder

Exclusion Criteria:

* any contraindication for MRI (orthodontia, vascular stent, metallic ear tubes, metal implants, piercings, etc.)
* neurological disorder, psychiatric disorder, or any major sensory deficit not associated with eating disorders or OCD (blindness, head trauma, bipolar disorder, seizure disorder, etc.)
* pregnancy
* below 85% of ideal body weight

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent females ages 12-19 drawn from clinic and community populations. With diagnosis of anorexia nervosa or obsessive-compulsive disorder or no psychiatric diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-01; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Brain activity related to set shifting | Baseline
Brain activity related to global vs. local processing | Baseline
Brain activity related to reward | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cara Bohon, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States